CLINICAL TRIAL: NCT03217097
Title: MGMT-NET: O6-methylguanine-DNA Methyltransferase (MGMT) Status in Neuroendocrine Tumors: Predictive Factor of Response to Alkylating Agents
Acronym: MGMT-NET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL17_0284
Record Dates: First submitted 2017-07-12; First posted 2017-07-13 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2022-11

CONDITIONS: Neuroendocrine Tumors
Keywords: Neuroendocrine tumors; Methylation MGMT status; Alkylating agents; Oxaliplatin
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Unmethylated MGMT NET - OX (Experimental): Patients with unmethylated MGMT NET will be randomly assigned (1:1) to either the alkylating-based chemotherapy arm or to the oxaliplatin-based chemotherapy arm.
  The "oxaliplatin-based" group will receive gemox (gemcitabine-oxaliplatin, 1x/2 week); alternatively folfox (5 fluorouracil-leucovorin-oxaliplatin, 1x/2 week) or capox (capecitabine-oxaliplatin, 1x/3 week).
  Interventions: Drug: Oxaliplatin-based chemotherapy
- Unmethylated MGMT NET - ALKY (Active Comparator): Patients with unmethylated MGMT NET will be randomly assigned (1:1) to either the alkylating-based chemotherapy arm or to the oxaliplatin-based chemotherapy arm.
  The "alkylating-based" group will receive CapTem regimen (capecitabine and temozolomide, /4 week), alternatively LV5FU2 (folinic acid-5 fluorouracil)-dacarbazine (1x/2 week) or LV5FU2 (folinic acid-5-fluorouracil)-streptozotocine (1x/2 week).
  Interventions: Drug: Alkylating-based chemotherapy
- Methylated MGMT NET - OX (Experimental): Patients with methylated MGMT NET will be randomly assigned (2:1) to either the alkylating-based chemotherapy arm or to the oxaliplatin-based chemotherapy arm.
  The "oxaliplatin-based" group will receive gemox (gemcitabine-oxaliplatin, 1x/2 week); alternatively folfox (5 fluorouracil-leucovorin-oxaliplatin, 1x/2 week) or capox (capecitabine-oxaliplatin, 1x/3 week).
  Interventions: Drug: Oxaliplatin-based chemotherapy
- Methylated MGMT NET - ALKY (Active Comparator): Patients with methylated MGMT NET will be randomly assigned (2:1) to either the alkylating-based chemotherapy arm or to the oxaliplatin-based chemotherapy arm.
  The "alkylating-based" group will receive CapTem regimen (capecitabine and temozolomide, /4 week), alternatively LV5FU2 (folinic acid-5 fluorouracil)-dacarbazine (1x/2 week) or LV5FU2 (folinic acid-5-fluorouracil)-streptozotocine (1x/2 week).
  Interventions: Drug: Alkylating-based chemotherapy

INTERVENTIONS:
Drug: Oxaliplatin-based chemotherapy — The "oxaliplatin-based" group will receive gemox (gemcitabine-oxaliplatin, 1x/2 week); alternatively folfox (5 fluorouracil-leucovorin-oxaliplatin, 1x/2 week) or capox (capecitabine-oxaliplatin, 1x/3 week).
  Arms: Methylated MGMT NET - OX; Unmethylated MGMT NET - OX
Drug: Alkylating-based chemotherapy — The "alkylating-based" group will receive CapTem regimen (capecitabine and temozolomide, /4 week), alternatively LV5FU2 (folinic acid-5 fluorouracil)-dacarbazine (1x/2 week) or LV5FU2 (folinic acid-5-fluorouracil)-streptozotocine (1x/2 week).
  Arms: Methylated MGMT NET - ALKY; Unmethylated MGMT NET - ALKY

SUMMARY:
Neuroendocrine tumors (NET) are rare but their incidence is growing. Alkylating agents (ALKY) are one of the main systemic treatments used, at least for advanced duodeno-pancreatic NETs, with a response rate of 30 to 40% and a median progression-free survival of 4 to 18 months. Chemotherapy is one of the few therapeutic weapons, along with everolimus, somatostatin analogs, and metabolic radiotherapy, for lung NETs, called typical and atypical carcinoids, even if the level of proof of efficacy for these treatments is lower than for duodeno-pancreatic NETs. Considering the available retrospective data, O6-Methylguanine-DNA methyltransferase (MGMT) appears to be a predictive factor of the response to ALKY. Oxaliplatin (OX) has demonstrated an interesting activity, with response rates between 17% and 30%. In a first retrospective study we showed that Gemox is effective in NET, and more recently that its activity is similar to that of ALKYs, but without being influenced by the MGMT status. Prospective studies are needed but our data suggests that ALKY should be offered first to patients with methylated MGMT tumors while Oxaliplatin-based chemotherapy should be offered first to patients with unmethylated MGMT tumors.

In this project, we wish to evaluate the contribution of the MGMT methylation, evaluated in the tumor, in predicting the Objective Response (OR) in patients treated with ALKY and to evaluate a treatment with alkylating agents versus Oxaliplatin in patients with a duodeno-pancreatic or lung or unknown primitive NET.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years;
* Patient presenting well-differentiated advanced grade 1-3 (locally/metastatic) duodeno-pancreatic or thoracic (lung or thymus) or unknown primitive NETs, not curable with surgery.
* Patients must have measurable disease using the RECIST v1.1 criteria;
* Indication for cytotoxic systemic chemotherapy validated by the dedicated Multidisciplinary Tumor Board;
* MRI or TAP CT scan with contrast agents within 4 weeks +/- 1 week before beginning of treatment;
* Tumor tissue available (fresh frozen or paraffin-embedded) in order to search for the methyl guanine methyltransferase (MGMT) status;
* Patients with childbearing potential should use effective contraception during the study and the following 6 months;
* Covered by a Healthcare System where applicable, and/or in compliance with the recommendations of the national laws in force relating to biomedical research;
* Subject able to understand and willing to sign a written informed consent document;
* Signed written informed consent obtained prior to any study-specific screening procedures.

Previous treatments such as surgery, radiofrequency ablation, transarterial liver embolization, somatostatin analogs, interferon, everolimus or other targeted therapy, peptide receptor radionuclide treatment (PRRT) and chemotherapy (platin-etoposide, folfiri, paclitaxel or docetaxel) are allowed.

Exclusion Criteria:

* Previous chemotherapy using Oxaliplatin or ALKY (streptozotocin, dacarbazin or temozolomide). Other chemotherapy (platin-etoposide, folfiri, paclitaxel or docetaxel) are allowed;
* Pregnant or breastfeeding;
* Men and women of childbearing age potential not using medically accepted contraceptive measures, as judged by the investigator;
* Contraindication to any drug contained in the chemotherapy regimen;
* Any significant disease which, in the investigator's opinion, excludes the patient from the study;
* Under any administrative or legal supervision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-04-25 (Actual)

PRIMARY OUTCOMES:
Objective Response (OR) in patients treated with alkylating-based chemotherapy | 3 months
  Objective Response (OR) in NETs patients treated with alkylating-based chemotherapy according to O6-Methyl guanine methyltransferase (MGMT) methylation status. The evaluation of OR is evaluation of complete response (CR) or partial response (PR) assessed by CT scan TAP or MRI with injection using the RECIST v1.1 criteria by centralized reading carried out by an expert radiologist blinded to the results of the MGMT methylation (methylated or un-methylated).

SECONDARY OUTCOMES:
Objective Response (OR) in patients treated with oxaliplatin-based chemotherapy | 3 months
  Objective Response (OR) in NETs patients treated with oxaliplatin-based chemotherapy according to O6-Methyl guanine methyltransferase (MGMT) methylation status. The evaluation of OR is evaluation of complete response (CR) or partial response (PR) assessed by CT scan TAP or MRI with injection using the RECIST v1.1 criteria by centralized reading carried out by an expert radiologist blinded to the results of the MGMT methylation (methylated or un-methylated).
Progression Free Survival (PFS) in patients treated with alkylating-based chemotherapy | 3 months
  Progression Free Survival (PFS) in patients treated with alkylating-based chemotherapy according to MGMT methylation status. Progression Free Survival (PFS) is defined as the time from random assignment in a clinical trial to disease progression (assessed by CT scan TAP or MRI with injection, using the RECIST v1.1 criteria by centralized reading carried out by an expert radiologist blinded to the results of the MGMT methylation) or death from any cause.
Progression Free Survival (PFS) in patients treated with oxaliplatin-based chemotherapy | 3 months
  Progression Free Survival (PFS) in patients treated with oxaliplatin-based chemotherapy according to MGMT methylation status. Progression Free Survival (PFS) is defined as the time from random assignment in a clinical trial to disease progression (assessed by CT scan TAP or MRI with injection, using the RECIST v1.1 criteria by centralized reading carried out by an expert radiologist blinded to the results of the MGMT methylation) or death from any cause.
Overall Survival (OS) in patients treated with alkylating-based chemotherapy | 3 months
  Overall Survival (OS) in patients treated with alkylating-based chemotherapy according to MGMT methylation status. Overall Survival (OS) is defined as the time from random assignment to the date of death due to any cause, or to the date of censoring at the last time the subject was known to be alive in intention-to-treat populations
Overall Survival (OS) in patients treated with oxaliplatin-based chemotherapy | 3 months
  Overall Survival (OS) in patients treated with oxaliplatin-based chemotherapy according to MGMT methylation status. Overall Survival (OS) is defined as the time from random assignment to the date of death due to any cause, or to the date of censoring at the last time the subject was known to be alive in intention-to-treat populations
Objective Response (OR) assessed by immunochemistry on tissue | 3 months
  Objective Response (OR) at 3 months assessed by RECIST v1.1 criteria in patients with unmethylated MGMT NETs and in patients with methylated MGMT NETs evaluated with immunochemistry (IHC) on tissue

CONTACTS AND LOCATIONS:
Locations (19):
- France (19):
  - Hôpital Sud - CHU Amiens, Amiens
  - CHU d'Angers, Angers
  - Hôpital Estaing, CHU de Clermont-Ferrand, Clermont-Ferrand
  - Hôpital Beaujon - APHP, Clichy
  - Hôpital François Mitterrand - CHU Dijon Bourgogne, Dijon
  - Centre Oscar Lambret, Lille
  - Hôpital Claude Hurriet - CHRU Lille, Lille
  - Hôpital Edouard Herriot - Hospices Civils de Lyon, Lyon
  - Hôpital Privé Jean Mermoz, Lyon
  - Institut Paoli Calmettes, Marseille
  - Hôpital Saint Louis - APHP, Paris
  - Hôpital Cochin - APHP, Paris
  - CH Annecy Genevois, Pringy
  - Hôpital Robert Debré - CHU Reims, Reims
  - Hôpital Nord - CHU Saint Etienne, Saint-Priest-en-Jarez
  - Institut de Cancérologie de la Loire, Saint-Priest-en-Jarez
  - Hôpital Rangueil - CHU Toulouse, Toulouse
  - Hôpital Trousseau - CHU Tours, Tours
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Result] Lemelin A, Barritault M, Hervieu V, Payen L, Peron J, Couvelard A, Cros J, Scoazec JY, Bin S, Villeneuve L, Lombard-Bohas C, Walter T; MGMT-NET investigators. O6-methylguanine-DNA methyltransferase (MGMT) status in neuroendocrine tumors: a randomized phase II study (MGMT-NET). Dig Liver Dis. 2019 Apr;51(4):595-599. doi: 10.1016/j.dld.2019.02.001. Epub 2019 Feb 14. PMID 30824408
- [Result] Walter T, Lecomte T, Hadoux J, Niccoli P, Saban-Roche L, Gaye E, Guimbaud R, Baconnier M, Hautefeuille V, Do Cao C, Petorin C, Hentic O, Perrier M, Aparicio T, Scoazec JY, Bonjour M, Gibert B, Hervieu V, Poncet D, Barritault M, Gerard L, Durand A; "Groupe d'etude des tumeurs endocrines (GTE)" and the French ENDOCAN-RENATEN network. Oxaliplatin-Based Versus Alkylating Agent in Neuroendocrine Tumors According to the O6-Methylguanine-DNA Methyltransferase Status: A Randomized Phase II Study (MGMT-NET). J Clin Oncol. 2025 Mar 10;43(8):960-971. doi: 10.1200/JCO.23.02724. Epub 2024 Nov 25. PMID 39586038